CLINICAL TRIAL: NCT02203201
Title: Diagnostic Significance of Positive Anti-endomysium Antibodies in the Culture Medium of the Intestinal Biopsies in Not-Celiac Wheat Sensitivity (NCWS)
Brief Title: Diagnostic Significance of Positive EmA Antibodies in the Duodenal Culture Medium of Not-Celiac Wheat Sensitivity (NCWS)
Acronym: NCWS
Status: Completed | Type: Observational
Sponsor: University of Palermo (Other)
Responsible Party: Principal Investigator, Pasquale Mansueto, Researcher, University of Palermo
Other Study IDs: ACPM04
Record Dates: First submitted 2014-06-14; First posted 2014-07-29 (Estimated); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Not-celiac Gluten Sensitivity
Keywords: Not-celiac gluten sensitivity; Celiac Disease; Gluten-free diet; EMA assay; Duodenal culture medium
MeSH Terms: conditions — Celiac Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Study group: NCWS patients who had showed a negative celiac disease serology and a Marsh 0-1 duodenal histology, but who had displayed a positive EmA assay in the culture medium of the duodenal biopsies (EmA-biopsy).
- Control group: NCWS patients with negative EmA-biopsy.

SUMMARY:
The most frequent diseases caused by wheat ingestion are T cell-mediated disorders, i.e. celiac disease and immunoglobulin E (IgE)-mediated allergic reactions. However, besides celiac disease and wheat allergy, there are cases of gluten reactions in which neither autoimmune nor IgE-mediated allergic mechanisms are involved. These are generally defined as GS or Not-celiac wheat sensitivity (NCWS). Typically, NCWS diagnosis is made by exclusion, and an elimination diet and an "open challenge" (i.e., the monitored reintroduction of gluten-containing foods) are most often used to evaluate whether health improves or worsen with the elimination or reintroduction of gluten in the diet, respectively. In some circumstances, it is very difficult to distinguish between NCWS and celiac disease. The presence of positive celiac disease specific serum antibodies (anti-tissue transglutaminase (anti-tTG), and anti-endomysium (EmAs) antibodies) is of paramount importance to pose the diagnosis. However, it is well known that the frequency of a positive serology is dependent by the severity of the intestinal damage. Consequently, patients with less severe histology damage (Marsh 1) can have negative serum antibodies. Previous studies had demonstrated that EmAs are produced by the intestinal lymphocytes and previous data from our group showed that EmAs assay in the culture medium of the intestinal biopsies has higher diagnostic accuracy than serum EmAs in diagnosis. Therefore, the aims of our study are to evaluate the clinical-serologic-histology course of NCWS patients, showing positive EmAs assay in the culture medium of the duodenal biopsies at the time of the first evaluation, and the adherence to a gluten-free diet in NCWS patients after a previous full evaluation and a NCWS diagnosis based on double-blinded placebo-controlled (DBPC) challenge.

DETAILED DESCRIPTION:
Gluten is the most important protein component of some grains, notably wheat, rye, and barley, which are the basis for a variety of wheat-derived alimentary products consumed throughout the world (bread, pasta, pizza etc). However the "engineering" of gluten-containing grains created the conditions for human diseases related to gluten exposure. These forms of gluten intolerance represent a heterogeneous set of conditions, including celiac disease, wheat allergy and gluten sensitivity (GS), that, combined, seems to affect about 10% of the general population.

The immune responsiveness to wheat antigens represents a complex process, and its establishment and maintenance are not completely elucidated. The most frequent diseases caused by wheat ingestion are T cell-mediated disorders, i.e. celiac disease and IgE-mediated allergic reactions. However, besides celiac disease and wheat allergy, there are cases of gluten reactions in which neither autoimmune nor IgE-mediated allergic mechanisms are involved. These are generally defined as GS or Not-celiac wheat sensitivity (NCWS), because it is not known what component of the cereals causes the symptoms. Some subjects, who experience symptoms when eating gluten-containing products and show improvement when following a gluten-free diet (GFD) may have NCWS instead of celiac disease or wheat allergy. NCWS patients are unable to tolerate gluten and develop an adverse reaction when eating gluten, that, usually, and differently from celiac disease, does not lead to small intestinal damage. Gastrointestinal symptoms in NCWS patients may resemble those associated with celiac disease, but the overall clinical picture is generally less severe.

Typically, NCWS diagnosis is made by exclusion, and an elimination diet and an "open challenge" (i.e., the monitored reintroduction of gluten-containing foods) are most often used to evaluate whether health improves or worsen with the elimination or reintroduction of gluten in the diet, respectively.

The frequency of NCWS is however still unknown, even though some studies indicated that it is higher than that of celiac disease; consequently, it is very probable that this condition have been undiagnosed and under-diagnosed by the physicians for a long time. However, it is very difficult, in some circumstances, to distinguish between NCWS and celiac disease. In fact, NCWS patients can show an intestinal histology characterized by intra-epithelial lymphocytosis (Marsh 1), a finding considered compatible with a celiac disease diagnosis. In this difficult, possible, celiac disease diagnosis, the presence of positive specific serum antibodies (anti-tTG and EmAs) is of paramount importance to pose the diagnosis. However, it is well known that the frequency of a positive serology is dependent by the severity of the intestinal damage. Consequently, celiac disease patients with less severe histology damage (Marsh 1) can have negative serum antibodies. Previous studies had demonstrated that EmAs are produced by the intestinal lymphocytes and previous data from our group showed that EmAs assay in the culture medium of the intestinal biopsies has higher diagnostic accuracy than serum EmAs in celiac disease diagnosis.

Therefore, this study has one major aim: 1. Evaluation of the clinical-serologic-histology course of NCWS patients showing positive EmAs assay in the culture medium of the duodenal biopsies at the time of the first evaluation; and one secondary aim: 2. Evaluation of the adherence to a GFD in NCWS patients after a previous full evaluation and a NCWS diagnosis based on double-blinded placebo-controlled (DBPC) challenge.

For our research, the investigators will select adult patients, both genders, affected with NCWS (i.e. with symptoms/signs which disappeared on gluten-free diet and worsen on a gluten containing diet, testing negative for celiac disease, [anti-tTG and EmAs negative, and with biopsy Marsh 0-1] and wheat allergy [serum specific IgE for wheat negative]).

The investigators will include exclusively patients who had been previously fully evaluated for suspected celiac disease in our Hospitals (Department of Internal Medicine, Giovanni Paolo II Hospital of Sciacca, Agrigento, and of Internal Medicine of the University of Palermo) from January 2002 to December 2012. In all patients NCWS diagnosis had been posed by means of a DBPC challenge with wheat flour. At the time of the first evaluation, gluten-free diet was not prescribed, but simply suggested, as these patients were not considered as suffering from celiac disease.

The investigators will recruit, as a study group, those NCWS patients who had showed a negative celiac disease serology and Marsh 0-1 duodenal histology, but who had displayed a positive EmAs assay in the culture medium of the duodenal biopsies (EmA-biopsy). As control group, NCWS patients with negative EmA-biopsy will be included.

The investigators will include at least one year before evaluated patients. At the time of the recruitment it will be evaluated both the adherence to the gluten-free diet, by means of a previously validated dietary form containing a printed list of the most common foods, and the symptoms score (Gastrointestinal Symptom Rating Scale, GSRS). Then, the investigators will re-evaluate the patients for a possible celiac disease diagnosis. Serum anti-tTG IgA and IgG, anti-deamidated peptides of gliadin (DPG) IgA and IgG, and anti-gliadin (AGA) IgA and IgG will be assayed. Duodenal biopsies will be taken for histological evaluation and for culture EmAs assay.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, both genders, with age between 18-65 years, that has been previously diagnosed as NCWS, according to a DBPC method
* Patients testing negative for celiac disease ( anti-tTG and EMA negative, and with biopsy Marsh 0-1) and wheat allergy (serum specific igE for wheat negative)
* Patients showed positive EmAs in the culture medium of the duodenal biopsies

Exclusion Criteria:

* Subjects diagnosed with celiac disease (positive anti-tTG and/or EMA, and positive histology, with Marsh 2 or above)
* Subjects diagnosed with wheat allergy (positive serum specific IgE for wheat)
* Subjects with Type 1 Diabetes
* Subjects with Inflammatory Bowel Diseases (Crohn's disease or ulcerative colitis)
* Subjects with Helicobacter pylori infection and other gastrointestinal infection
* Pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The investigators will include exclusively patients who had been previously fully evaluated for suspected celiac disease in our Hospitals (Department of Internal Medicine, Giovanni Paolo II Hospital of Sciacca, Agrigento, and of Internal Medicine of the University of Palermo) from January 2002 to December 2012. In all patients NCWS diagnosis had been posed by means of a double-blind placebo-controlled (DBPC) challenge with wheat flour.
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2016-10-01 (Actual); Study Completion 2020-06-01 (Actual)

PRIMARY OUTCOMES:
Changes in the intestinal histology of NCWS patients who tested positives for EmAs in the culture medium of the intestinal biopsies, at the time of the first evaluation. | At baseline and after at least one year since the initial NCWS diagnosis was posed.
  Intestinal histology re-evaluation after at least one year since the initial NCWS diagnosis was posed. Marsh classification will be adopted: change from baseline (1st evaluation) to 2nd evaluation.
  The above parameter will be evaluated taking into account whether the patients adhered or not to a wheat-free diet.

SECONDARY OUTCOMES:
Serum anti-tTG antibodies evaluation. | At baseline and after at least one year since the initial NCWS diagnosis was posed.
  Evaluation of changes in serum levels of anti-tTG antibodies after at least one year since the initial NCWS diagnosis was posed.
Serum DPG antibodies evaluation. | At baseline and after at least one year since the initial NCWS diagnosis was posed.
  Evaluation of changes in serum levels of DPG antibodies after at least one year since the initial NCWS diagnosis was posed.
Serum AGA evaluation. | At baseline and after at least one year since the initial NCWS diagnosis was posed.
  Evaluation of changes in serum levels of AGA after at least one year since the initial NCWS diagnosis was posed.
Adherence to a wheat-free diet | At baseline and after at least one year since the initial NCWS diagnosis was posed.
  Degree of adherence to a wheat-free diet since the initial diagnosis of NCWS was posed.
Symptoms/signs evaluation. | At baseline and after at least one year since the initial NCWS diagnosis was posed.
  The evaluation of changes in symptoms/signs will be made according to the score calculated on the basis of the Visual Analogue Scale since the initial diagnosis of NCWS was posed.

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Carroccio, MD, PhD, Study Director — University of Palermo; Pasquale Mansueto, MD, Principal Investigator — University of Palermo
Locations (2):
- Italy (2):
  - Department of Internal Medicine, Giovanni Paolo II Hospital of Sciacca, Sciacca, Agrigento
  - Department of Internal Medicine, University Hospital of Palermo, Palermo

REFERENCES:
- [Background] Carroccio A, Iacono G, Di Prima L, Pirrone G, Cavataio F, Ambrosiano G, Sciume C, Geraci G, Florena A, Teresi S, Barbaria F, Pepe I, Campisi G, Mansueto P, Soresi M, Di Fede G. Antiendomysium antibodies assay in the culture medium of intestinal mucosa: an accurate method for celiac disease diagnosis. Eur J Gastroenterol Hepatol. 2011 Nov;23(11):1018-23. doi: 10.1097/MEG.0b013e328349b8a5. PMID 21885984
- [Background] Carroccio A, Iacono G, D'Amico D, Cavataio F, Teresi S, Caruso C, Di PL, Colombo A, D'Arpa F, Florena A, Notarbartolo A, Montalto G. Production of anti-endomysial antibodies in cultured duodenal mucosa: usefulness in coeliac disease diagnosis. Scand J Gastroenterol. 2002 Jan;37(1):32-8. doi: 10.1080/003655202753387329. PMID 11843032